CLINICAL TRIAL: NCT02203084
Title: The Influence of Social Determinants and Access to Health Care on the Outcome of Children With Chronic Health Problems in British Columbia
Brief Title: Social Determinants in Chronic Disease in British Columbia
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Michael Seear, Principle Investigator, University of British Columbia
Other Study IDs: H14-01278
Record Dates: First submitted 2014-07-25; First posted 2014-07-29 (Estimated); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: Cystic Fibrosis; Diabetes Mellitus Type I; Chronic Renal Insufficiency
Keywords: Cystic Fibrosis; Diabetes Mellitus Type I; Chronic Renal Insufficiency; The influence of socioeconomic variables upon outcome in children with three chronic medical diseases.
MeSH Terms: conditions — Cystic Fibrosis; Diabetes Mellitus, Type 1; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Children with Chronic Medical Conditions: The Social Determinants Questionnaire will be administered to the three groups of children with chronic diseases (cystic fibrosis, diabetes mellitus type I, or chronic renal insufficiency). The questionnaire questions will be asked by a research assistant. Each participant will have the same general and background information questions then will have questions specific to their chronic medical condition.
  Interventions: Other: Social Determinants Questionnaire

INTERVENTIONS:
Other: Social Determinants Questionnaire — The questionnaire contains a general background information section common to all medical conditions. It then contains separate sections with medical condition specific questions.

SUMMARY:
Anyone who practices clinical medicine will understand that socially disadvantaged children will have worse health outcomes, no matter what the underlying condition might be. There is limited prospective data on the effects of social deprivation on children in BC and there is none concerning the effects of social deprivation on children with chronic diseases. In order to generate relevant data for those who manage children with chronic diseases in BC, the investigators wish to perform an observational study of the relationship between questionnaire-derived social variables and measured outcomes in children with cystic fibrosis, type 1 diabetes, and chronic kidney disease.

Our working hypothesis is that there is an association between social determinants of health (income, education, race) and health outcomes in children with cystic fibrosis, type 1 diabetes and chronic renal failure, that is independent of access to health care (assessed by distance to nearest specialty clinic and number of clinic visits in the last year).

DETAILED DESCRIPTION:
1. Cystic fibrosis (CF). Cystic fibrosis is a genetic condition that causes slowly progressive lung disease. It occurs in people of all social class so the disease itself is independent of social factors. There is considerable variation in the outcome of CF in different children. There are many potential causes for these differences but the available literature would suggest that a significant part of this variability is due to social factors. While there are no prospective clinical studies, the limited information from database reviews suggest that socially deprived children have significantly worse outcomes. In the US, children living in poverty are twice as likely to be underweight and over three times more likely to die (25). UK data is similar - disadvantaged children have worse growth parameters and lower lung function compared to richer children (26).
2. Type 1 diabetes (T1D). Type 1 diabetes is a multi-factorial disease. It is not an autosomal recessive disease like CF but genetic predisposition can be one of its predisposing features. As with the data on CF, socio-economic deprivation has been shown to have a significant adverse effect on outcome in type 1 diabetes. In the US, glycemic control amongst young adults was significantly worse amongst disadvantaged young adults (27). A retrospective review of New Zealand children with type 1 diabetes also showed that poor socio-economic status and Polynesian ethnicity were significantly associated with poor glycemic control and long term complications (28).
3. Chronic kidney disease (CKD). Chronic kidney disease may be due to congenital, acquired, or hereditary causes. Within all these groups, socioeconomic status, gender, and race may influence disease progression and outcomes. It has been shown in children with chronic kidney disease, primarily from the United States, that it was more common in low- and middle- income families to have an abnormal birth history such as prematurity, low birth weight or small for age which predisposes to the development of renal disease (29). In addition, blood pressure control and height deficits improve faster in children of families with higher income. In Canada, Aboriginals have a higher prevalence of severe chronic kidney disease and a 77% increased mortality risk (30,31) and a lower likelihood of nephrology clinic visits (32). Aboriginal children and young adults with chronic kidney disease are more likely to have glomerulonephritis as a cause of kidney disease compared to Caucasians and are more likely to reach end stage renal disease (33). In contrast, lower mortality risks are seen in East Asian and Indo Asian Canadian adults starting dialysis (34). There is still much to be studied on the influence of these various factors in renal health and disease.

STUDY DESIGN.

1. Study Objective. We wish to determine the influence of education, income, race and access to health care upon health outcomes in children with chronic diseases in British Columbia.
2. Justification. While the effects of social deprivation on health outcomes are commonly discussed, it is surprising how little prospective research there is to quantify the adverse effects of social inequity. There is limited prospective data on the effects of social deprivation on children in BC and there is none concerning the effects of social deprivation on children with chronic diseases. In order to generate firm data relevant for those who manage children with chronic diseases in BC, we wish to perform a cross sectional observational study of the relationship between social variables and outcome in children with cystic fibrosis, type 1 diabetes and chronic kidney disease.
3. General design. All families in the three clinics will initially be informed of the study by letter. When the child is due for regular follow-up assessment, the parents will be approached during the clinic visit and invited to join the study. Their participation will only involve the completion of a questionnaire. The research assistant will collect the data at interview and will subsequently (with parental permission) retrieve laboratory results from records of previous clinic visits to assess measured health trends over time. The study protocol does not add any further investigations other than the questionnaire. Apart from the variable time needed for parent information and consent, the questionnaire itself will require no more than about 30 minutes to complete.
4. Questionnaire. We will use a socio-economic assessment questions that we are already using in our study of quality of life in parents caring for children needing home ventilation. It is a conventional form assessing education level, employment, income, partnership status and ethnicity. This last is very important because of the poorer health outcomes already known to be associated with Aboriginal background. The proxy for access to health care will be distance to the main specialty clinic and number of visits in the last year.
5. Analysis. The relationship between socio-economic variables plus ethnicity and outcome will be examined using multiple linear regression analysis. In the absence of relevant literature, there are too many unknowns to allow any reliable form of power analysis or patient number calculation to be performed. One accepted 'rule of thumb' is that there should be at least 10 patients for each predictive variable in multiple linear regression analysis. We will concentrate on 6 to 8 of the main social factors and will try to enroll over 100 patients within each sub-specialty - enough to ensure 15 to 20 patient outcomes for each variable.

ELIGIBILITY:
Inclusion Criteria:

* Any individual who attends British Columbia Children's Hospital Ambulatory clinics in the following areas: cystic fibrosis, chronic kidney disease, or type 1 diabetes

Exclusion Criteria:

* Refusal to join the study
* Acute Medical Instability

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants will be sampled from the cystic fibrosis clinic (150) patients and the chronic kidney disease clinic (150 patients). For the larger type 1 diabetes clinic the sample will be purposefully stratified. Recruitment will be monitored to ensure adequate representation from all the health authorities in BC.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2014-09-01; Primary Completion 2017-06-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Level of glycosylated hemoglobin (HbA1C) | 1 year
  The level of glycosylated hemoglobin (HbA1C) is the conventional measure of glycemic control and will be used to assess the diabetic group. Data is measured every 3-6 months and will be collected from previous clinic visits. Measurements performed routinely at clinic visits. The monitoring results will be recorded but the study does not require or involve any testing other than tests associated with routine clinical practice.
Height/weight | 1 year
  Height/weight used to assess cystic fibrosis patients. Measurements performed routinely at clinic visits. The monitoring results will be recorded but the study does not require or involve any testing other than tests associated with routine clinical practice.
Lung Function Tests | 1 year
  Lung function tests used to assess cystic fibrosis patients. Measurements performed routinely at clinic visits. The monitoring results will be recorded but the study does not require or involve any testing other than tests associated with routine clinical practice.
Glomerular filtration rate (GFR) | 1 year
  GFR used to assess renal failure patients. Measurements performed routinely at clinic visits. The monitoring results will be recorded but the study does not require or involve any testing other than tests associated with routine clinical practice.
Albumin/creatinine ratio | 1 year
  Albumin/creatinine ratio used to assess renal failure patients. Measurements performed routinely at clinic visits. The monitoring results will be recorded but the study does not require or involve any testing other than tests associated with routine clinical practice.

CONTACTS AND LOCATIONS:
Overall Officials: Mike Seear, MD, Principal Investigator — British Columbia's Children's Hospital; Mike Seear, MD, Principal Investigator — BCCH
Locations (1):
- BC's Children's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Schechter MS, Shelton BJ, Margolis PA, Fitzsimmons SC. The association of socioeconomic status with outcomes in cystic fibrosis patients in the United States. Am J Respir Crit Care Med. 2001 May;163(6):1331-7. doi: 10.1164/ajrccm.163.6.9912100. PMID 11371397
- [Background] Taylor-Robinson DC, Smyth RL, Diggle PJ, Whitehead M. The effect of social deprivation on clinical outcomes and the use of treatments in the UK cystic fibrosis population: a longitudinal study. Lancet Respir Med. 2013 Apr;1(2):121-8. doi: 10.1016/S2213-2600(13)70002-X. Epub 2013 Jan 30. PMID 24429092
- [Background] Secrest AM, Costacou T, Gutelius B, Miller RG, Songer TJ, Orchard TJ. Associations between socioeconomic status and major complications in type 1 diabetes: the Pittsburgh epidemiology of diabetes complication (EDC) Study. Ann Epidemiol. 2011 May;21(5):374-81. doi: 10.1016/j.annepidem.2011.02.007. PMID 21458731
- [Background] Carter PJ, Cutfield WS, Hofman PL, Gunn AJ, Wilson DA, Reed PW, Jefferies C. Ethnicity and social deprivation independently influence metabolic control in children with type 1 diabetes. Diabetologia. 2008 Oct;51(10):1835-42. doi: 10.1007/s00125-008-1106-9. Epub 2008 Aug 5. PMID 18679654
- [Background] Hidalgo G, Ng DK, Moxey-Mims M, Minnick ML, Blydt-Hansen T, Warady BA, Furth SL. Association of income level with kidney disease severity and progression among children and adolescents with CKD: a report from the Chronic Kidney Disease in Children (CKiD) Study. Am J Kidney Dis. 2013 Dec;62(6):1087-94. doi: 10.1053/j.ajkd.2013.06.013. Epub 2013 Aug 7. PMID 23932090
- [Background] Gao S, Manns BJ, Culleton BF, Tonelli M, Quan H, Crowshoe L, Ghali WA, Svenson LW, Hemmelgarn BR; Alberta Kidney Disease Network. Prevalence of chronic kidney disease and survival among aboriginal people. J Am Soc Nephrol. 2007 Nov;18(11):2953-9. doi: 10.1681/ASN.2007030360. Epub 2007 Oct 17. PMID 17942955
- [Background] Bulloch B, Postl BD, Ogborn MR. Excess prevalence of non diabetic renal disease in native American children in Manitoba. Pediatr Nephrol. 1996 Dec;10(6):702-4. doi: 10.1007/s004670050193. PMID 8971883
- [Background] Gao S, Manns BJ, Culleton BF, Tonelli M, Quan H, Crowshoe L, Ghali WA, Svenson LW, Ahmed S, Hemmelgarn BR; Alberta Kidney Disease Network. Access to health care among status Aboriginal people with chronic kidney disease. CMAJ. 2008 Nov 4;179(10):1007-12. doi: 10.1503/cmaj.080063. PMID 18981441
- [Background] Samuel SM, Foster BJ, Hemmelgarn BR, Nettel-Aguirre A, Crowshoe L, Alexander RT, Soo A, Tonelli MA; Pediatric Renal Outcomes Canada Group. Incidence and causes of end-stage renal disease among Aboriginal children and young adults. CMAJ. 2012 Oct 2;184(14):E758-64. doi: 10.1503/cmaj.120427. Epub 2012 Aug 27. PMID 22927509
- [Background] Yeates K. Health disparities in renal disease in Canada. Semin Nephrol. 2010 Jan;30(1):12-8. doi: 10.1016/j.semnephrol.2009.10.014. PMID 20116643